CLINICAL TRIAL: NCT06504940
Title: Orelabrutinib Combined With BR/G Followed by Orelabrutinib Maintenance Therapy for Newly Diagnosed Marginal Zone Lymphoma (MZL): A Prospective ,Multicenter, Clinical Study
Brief Title: Optimize Study - Orelabrutinib Combined With BR/G in Untreated Marginal Zone Lymphoma (MZL)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT20240202
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Marginal Zone Lymphoma
Keywords: orebrutinib; BTKi; Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Bendamustine Hydrochloride; Rituximab; obinutuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): For individuals under 70 years of age with good fitness,
  Interventions: Drug: Orelabrutinib combined with bendamustine and rituximab
- Cohort B (Experimental): For individuals aged 70 or older or those under 70 years with poor fitness
  Interventions: Drug: Orelabrutinib combined with obinutuzumab

INTERVENTIONS:
Drug: Orelabrutinib combined with bendamustine and rituximab — they will receive three cycles of Orelabrutinib combined with bendamustine and rituximab (BR: bendamustine 70mg/m^2 on days 1-2; rituximab 375mg/m^2 on day 0). Patients achieving PR or better will enter the Orelabrutinib monotherapy maintenance phase (up to 21 cycles, each cycle 28 days).
  Arms: Cohort A
Drug: Orelabrutinib combined with obinutuzumab — they will receive six cycles of Orelabrutinib combined with obinutuzumab (G 1000mg iv on days 1, 8, 15 of cycle 1, and day 1 of cycles 2-6; Orelabrutinib 150mg once daily). Patients achieving PR or better will enter the Orelabrutinib monotherapy maintenance phase (up to 18 cycles, each cycle 28 days ).
  Arms: Cohort B

SUMMARY:
This is a multi-center, prospective cohort study. The main purpose of Cohort A is to evaluate the efficacy and safety of Orelabrutinib combined with BR (bendamustine and rituximab) for previously untreated young patients with MZL; the purpose of Cohort B is to assess the efficacy and safety of Orelabrutinib combined with G (Obinutuzumab) followed by Orelabrutinib maintenance therapy for previously untreated elderly patients with MZL.

DETAILED DESCRIPTION:
Marginal Zone Lymphoma (MZL) is a group of B-cell malignancies believed to originate from B lymphocytes, typically found in the marginal zones of lymphoid follicles in the spleen, lymph nodes, and mucosa-associated lymphoid tissues. Currently, there is no unified, high-level evidence-based treatment plan for previously untreated MZL. Exploring more effective, low-toxicity treatment plans for MZL patients is a scientifically valuable and clinically significant attempt. With the development of new drugs, new drug regimens have become prominent in the treatment of MZL, and there is an increasing amount of research data on BTK inhibitors in the field of MZL. The BTK inhibitor Orelabrutinib has shown good efficacy in MZL and has been approved by the NMPA for the treatment of MZL in patients who have received at least one prior treatment.

This study is a multi-center, prospective cohort clinical study for previously untreated MZL. Cohort A: For individuals under 70 years of age with good fitness, they will receive three cycles of Orelabrutinib combined with bendamustine and rituximab (BR: bendamustine 70mg/m^2 on days 1-2; rituximab 375mg/m^2 on day 0). Patients achieving PR or better will enter the Orelabrutinib monotherapy maintenance phase (up to 21 cycles, each cycle 28 days). Cohort B: For individuals aged 70 or older or those under 70 years with poor fitness, they will receive six cycles of Orelabrutinib combined with obinutuzumab (G 1000mg iv on days 1, 8, 15 of cycle 1, and day 1 of cycles 2-6; Orelabrutinib 150mg once daily). Patients achieving PR or better will enter the Orelabrutinib monotherapy maintenance phase (up to 18 cycles, each cycle 28 days ).

ELIGIBILITY:
Inclusion Criteria:

1. For Cohort A: Age 18-70 years, physical condition assessed by a physician as suitable for chemotherapy; for Cohort B: Age 70 or older or under 70 years of age assessed by a physician as unsuitable for chemotherapy.
2. Gender is not limited.
3. Confirmed by histopathology, marginal zone lymphoma including MALT, SMZL, NMZL.
4. Progression, recurrence after local treatment, or unsuitable for local treatment (local treatments include surgery, radiotherapy, Helicobacter pylori treatment, hepatitis C treatment).
5. ECOG performance score 0-3 points (if the score is 3 points, the physician needs to assess that the deterioration of physical condition is mainly due to tumor burden).
6. Indications for treatment (with B symptoms, blood cell decline, bleeding, large mass, rapid progression of tumors, etc.).
7. Major organ functions meet the following criteria: a) Complete blood count: Absolute neutrophil count ≥1.5×10^9/L, platelets ≥75×10^9/L, hemoglobin ≥75g/L; if accompanied by bone marrow involvement, absolute neutrophil count ≥1.0×10^9/L, platelets ≥50×10^9/L, hemoglobin ≥50g/L. b) Blood biochemistry: Total bilirubin ≤1.5 times the upper limit of normal (ULN), AST or ALT ≤2 times ULN; serum creatinine ≤1.5 times ULN; serum amylase ≤ULN. c) Coagulation function: International normalized ratio (INR) ≤1.5 times ULN.
8. Life expectancy ≥3 months.
9. Voluntarily sign a written informed consent form before the trial screening.

Exclusion Criteria:

1. Currently or previously have other malignant tumors, unless radical treatment has been performed and there is evidence of no recurrence or metastasis within the last 5 years.
2. Lymphoma involving the central nervous system or transformation to a higher grade.
3. Have uncontrollable or significant cardiovascular diseases, including: a) Within 6 months before the first administration of the study drug, there is a history of New York Heart Association (NYHA) class II or above congestive heart failure, unstable angina, myocardial infarction, or arrhythmias requiring treatment at the time of screening, with a left ventricular ejection fraction (LVEF) <50%. b) Primary cardiomyopathy (such as dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, unclassified cardiomyopathy). c) A history of clinically significant QTc interval prolongation, or a QTc interval >470ms in females and >450ms in males during the screening period. d) Symptomatic or medication-requiring coronary artery heart disease subjects. e) Subjects with uncontrollable hypertension (despite lifestyle improvements and the use of reasonable, tolerable, and adequate doses of three or more antihypertensive drugs, including diuretics, for more than 1 month, blood pressure is still not at the standard, or it is only effectively controlled when taking four or more antihypertensive drugs).
4. Active bleeding within 2 months before screening, or currently taking anticoagulant drugs, or the investigator believes there is a clear bleeding tendency.
5. History of deep vein thrombosis or pulmonary embolism within the past six months.
6. Clinically significant gastrointestinal abnormalities that may affect the intake, transport, or absorption of drugs (such as inability to swallow, chronic diarrhea, intestinal obstruction), or subjects who have undergone total gastrectomy.
7. History of organ transplantation or allogeneic bone marrow transplantation.
8. Major surgery within 6 weeks before screening or minor surgery within 2 weeks before screening. Major surgery is surgery that uses general anesthesia, but endoscopic examinations for diagnostic purposes are not considered major surgery. Insertion of vascular access devices will be exempt from this exclusion criterion.
9. Active infection or uncontrolled HBV (positive for HBsAg and/or HBcAb with positive HBV DNA titer), positive for HCV Ab, HIV/AIDS, or other serious infectious diseases; define active infection.
10. Subjects currently with pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, etc., that seriously affect lung function.
11. Previously treated with BTK, BCR pathway inhibitors (such as PI3K, Syk), and BCL-2 inhibitors.
12. Pregnant, breastfeeding women, and subjects of childbearing age who are unwilling to take contraceptive measures.
13. Need to continuously take drugs with moderate to severe inhibitory effects on cytochrome P450 CYP3A or strong inductive effects.
14. Other situations deemed unsuitable for participating in this trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2027-07-08 (Estimated); Study Completion 2029-07-08 (Estimated)

PRIMARY OUTCOMES:
Cohort A: The incidence of grade 3-5 adverse events (AEs) | From the first administration of the drug to one month after the completion of induction therapy.
  Adverse events will be graded by the investigator according to the NCI-CTCAE Version 5.0.
Cohort A:the complete response rate (CRR) | At 12 months.
  CRR is defined as the proportion of patients with a response of CR
Cohort B: The 2-year progression-free survival (PFS) rate. | From date of signing the informed consent until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years]
  Progression free survival (PFS) is defined as the time from registration to the first occurrence of progression or relapse as assessed by the investigator, or death from any cause. PFS for patients without disease progression, relapse, or death will be censored at the time of the last tumor assessment.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  The ORR is defined as the proportion of patients with a response of CR or PR
The 2-year overall survival (OS) rate | From date of signing the informed consent until the date of death from any cause, whichever came first, assessed up to 2 years
  Overall survival is defined as the period from the induction registration to death from any cause. Patients who have not died until the time of the analysis will be censored at their last contact date.
The 2-year progression-free survival (PFS) rate. | From date of signing the informed consent until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Progression free survival (PFS) is defined as the time from registration to the first occurrence of progression or relapse as assessed by the investigator, or death from any cause. PFS for patients without disease progression, relapse, or death will be censored at the time of the last tumor assessment.
Duration of response | Up to 2 years
  Duration of response as defined as the period from the first response (at least PR) to treatment until evidence of disease progression, relapse or death of any cause. Patients alive without progression and relapse will be censored at the latest tumor assessment date or the stopping date.
TTR | Up to 2 years
  TTR is defined as the time from registration to the first response.
The frequency of grade 3-5 AEs | From the first drug administration to one month after the end of treatment.
  Adverse events will be graded by the investigator according to the NCI-CTCAE Version 5.0.
The occurrence of adverse events and serious adverse events | From the first drug administration to one month after the end of treatment.
  7. Adverse events will be graded by the investigator according to the NCI-CTCAE Version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital ，Zhejiang University School of Medicine, Hangzhou, Zhejiang, China